CLINICAL TRIAL: NCT05255601
Title: A Phase 1/2 Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Relatlimab Plus Nivolumab in Pediatric and Young Adult Participants With Recurrent or Refractory Classical Hodgkin Lymphoma and Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Preliminary Efficacy of Relatlimab Plus Nivolumab in Pediatric and Young Adults With Hodgkin and Non-Hodgkin Lymphoma
Acronym: RELATIVITY-069
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA224-069; 2023-503715-14 (Other: EU CTR); U1111-1264-4062 (Registry Identifier: WHO)
Expanded Access: NCT05170685 (No longer available)
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Pediatric; Lymphoma, Non-Hodgkin; Hodgkin Disease; Relatlimab; Nivolumab; Lymphocyte Activation Gene-3; Lymphoma, Large B-Cell, Diffuse; Primary Mediastinal B-cell Lymphoma; Lymphoma, Large-Cell, Anaplastic; Burkitt lymphoma; Lymphoblastic lymphoma; NK/ T-cell lymphoma; Peripheral T-cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relatlimab + Nivolumab (Experimental)
  Interventions: Drug: Relatlimab; Drug: Nivolumab

INTERVENTIONS:
Drug: Relatlimab — Specified Dose on Specified Days
  Other Names: BMS-986016
Drug: Nivolumab — Specified Dose on Specified Days
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to assess the safety, tolerability, drug levels, and preliminary efficacy of relatlimab plus nivolumab in pediatric and young adult participants with recurrent or refractory classical Hodgkin lymphoma and non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants with pathologically confirmed high-risk R/R cHL, after non-response to or failure of 1or more lines of standard therapy.
* Participants with pathologically confirmed R/R NHL after non-response to or failure of 1or more lines of standard therapy, including, but not limited to, R/R primary mediastinal B-cell lymphoma, diffuse large B-cell lymphoma (DLBCL), mediastinal gray zone lymphoma (MGZL), anaplastic large cell lymphoma (ALCL), or peripheral T-cell lymphoma (PTCL).
* Participants with pathologically confirmed R/R NHL after non-response to or failure of 2 or more lines of standard therapy, including Burkitt lymphoma (blast count <25% malignant Burkitt cells and/or per the investigator's clinical assessment of risk status), lymphoblastic lymphoma (blast count < 25% of marrow nucleated cells and/or per the investigator's clinical assessment of risk status), NK/T-cell lymphoma (nasal and non-nasal NK/T-cell lymphoma subtypes, but not aggressive NK/T-cell leukemia/lymphoma subtype).
* The participant's current disease state must be R/R to standard therapy.
* Participants must have measurable PET positive disease in both cHL and NHL cohorts.

Exclusion Criteria:

* Primary CNS lymphoma of the brain or spinal cord, and secondary CNS lymphoma (ie, from systemic non-Hodgkin lymphoma) involving the brain, spinal cord, or with leptomeningeal seeding.
* Prior treatment with an anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways, with the exception of anti-PD(L)-1 targeted therapies.
* Prior treatment with lymphocyte activation gene-3 (LAG-3)-targeted agents.
* Participants with clinically significant systemic illnesses unrelated to the cancer as judged by the investigators, which would compromise the participant's ability to tolerate the study treatment.
* Participants with autoimmune disease.
* Prior allogeneic bone marrow transplantation.

Other protocol-defined inclusion/exclusion criteria apply

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2028-07-05 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 135 days following last dose
  DLT evaluation window is 4 weeks from start of treatment. Safety evaluation will continue up to 135 days following last dose.
Maximum tolerated dose or Recommended phase 2 dose (MTD/RP2D) | Up to 135 days following last dose
Number of participants with Adverse Events (AEs) | Up to 135 days following last dose
Number of participants with serious adverse events (SAEs) | Up to 135 days following last dose
Number of participants with AEs leading to discontinuation | Up to 135 days following last dose
Number of deaths | Up to 2 years from the last treatment of last participant
Number of participants with clinical laboratory abnormalities | Up to 135 days following last dose
Maximum observed plasma concentration (Cmax) | Up to 96 weeks
Trough observed concentration (Ctrough) | Up to 96 weeks
Time of maximum observed plasma concentration (Tmax) | Up to 96 weeks
Area Under the Curve within a dosing interval (AUC(TAU)) | Up to 96 weeks
Complete Metabolic Response (CMR) Rate defined as the proportion of all response-evaluable participants who achieve the best response of CMR using Lugano 2014 criteria | Up to 2 years from the last treatment of last participant

SECONDARY OUTCOMES:
Number of participants with AEs | Up to 135 days following last dose
Number of participants with SAEs | Up to 135 days following last dose
Number of participants with AEs leading to discontinuation | Up to 135 days following last dose
Number of deaths | Up to 2 years from the last treatment of last participant
Number of participants with clinical laboratory abnormalities | Up to 135 days following last dose
Overall Response Rate (ORR) defined as the proportion of all response- evaluable participants who achieve a best response of CMR or partial metabolic response (PMR) using the Lugano 2014 classification | Up to 2 years from the last treatment of last participant

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (76):
- United States (22):
  - Local Institution - 0077, Birmingham, Alabama
  - Local Institution - 0024, Phoenix, Arizona
  - Local Institution - 0035, Palo Alto, California
  - Local Institution - 0032, New Haven, Connecticut
  - Local Institution - 0061, Wilmington, Delaware
  - Local Institution - 0066, Fort Myers, Florida
  - Local Institution - 0017, Orlando, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Local Institution - 0073, Baltimore, Maryland
  - Local Institution - 0025, Minneapolis, Minnesota
  - Local Institution - 0020, Jackson, Mississippi
  - Local Institution - 0012, St Louis, Missouri
  - Local Institution - 0071, Hackensack, New Jersey
  - Local Institution - 0060, New York, New York
  - Local Institution - 0016, The Bronx, New York
  - Local Institution - 0059, Valhalla, New York
  - Local Institution - 0019, Hershey, Pennsylvania
  - Local Institution - 0014, Nashville, Tennessee
  - Local Institution - 0029, Austin, Texas
  - Local Institution - 0026, San Antonio, Texas
  - Local Institution - 0076, Norfolk, Virginia
  - UW Health - American Family Children's Hospital Pediatric Bone Marrow Transplant Clinic, Madison, Wisconsin
- Australia (3):
  - Local Institution - 0037, Randwick, New South Wales
  - Royal Childrens Hospital RCH - Queensland Childrens Hospital, South Brisbane, Queensland
  - Local Institution - 0042, Nedlands, Western Australia
- France (11):
  - CHU dAngers - Pole Pediatrie, Angers, Angers Cedex 9
  - Groupe Hospitalier Pellegrin - Hopital des enfants, Bordeaux
  - Local Institution - 0033, Caen
  - Local Institution - 0067, La Tronche
  - Institut d Hematologie et d Oncologie Pediatriques, Lyon
  - Local Institution - 0034, Marseille
  - Centre Hospitalier Universitaire de Montpellier CHU Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Armand-Trousseau, Paris
  - Assistance Publique-Hopitaux de Paris AP-HP - Hopital Universitaire Robert-Debre, Paris
  - Local Institution - 0022, Rennes
  - CHRU de Strasbourg-Hopital de Hautepierre, Strasbourg
- Germany (6):
  - Local Institution - 0056, Aachen
  - Local Institution - 0015, Berlin
  - Local Institution - 0028, Giessen
  - Local Institution - 0036, Hamburg
  - Local Institution - 0051, Munich
  - Local Institution - 0008, Münster
- Italy (12):
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan, Milano
  - Local Institution - 0010, Aviano
  - Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Local Institution - 0040, Florence
  - Local Institution - 0005, Genoa
  - Local Institution - 0070, Milan
  - Fondazione MBBM - Clinica Pediatrica, Monza
  - Local Institution - 0013, Napoli
  - Azienda Ospedale Universita Padova, Padua
  - Local Institution - 0041, Pavia
  - Local Institution - 0002, Roma
  - Local Institution - 0004, Turin
- Princess Maxima Center for pediatric oncology, Utrecht, Netherlands
- Spain (13):
  - Local Institution - 0069, Esplugues de Llobregat, Barcelona
  - Local Institution - 0046, Barcelona
  - Local Institution - 0009, Barcelona
  - Local Institution - 0030, Madrid
  - Local Institution - 0058, Madrid
  - Local Institution - 0044, Madrid
  - Local Institution - 0055, Madrid
  - Local Institution - 0045, Madrid
  - Local Institution - 0062, Pamplona
  - Local Institution - 0011, Santander
  - Local Institution - 0038, Seville
  - Local Institution - 0023, Seville
  - Local Institution - 0049, Valencia
- United Kingdom (8):
  - Local Institution - 0075, Cambridge, Cambridgeshire
  - Local Institution - 0074, Liverpool, England
  - Local Institution - 0054, London, Londonderry
  - Local Institution - 0003, Nottingham, Nottinghamshire
  - Local Institution - 0050, Bristol, Somerset
  - Local Institution - 0068, Newcastle upon Tyne, Tyne and Wear
  - Local Institution - 0031, Birmingham, West Midlands
  - Local Institution - 0053, London

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05255601.html